CLINICAL TRIAL: NCT06685068
Title: A Phase 1/2 Study of GEN1286 in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1286-01; CTR20250215 (Registry Identifier: China Drug Trials); PRO1286-001 (Other: Sponsor identifier)
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: No randomization will be performed in Part A (dose escalation- sequential assignment). In Part B (tumor-specific expansion- parallel assignment), participants in each cohort will be randomized with a 1:1 ratio to receive one of the expansion doses of GEN1286.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GEN1286 (Experimental)
  Interventions: Drug: GEN1286

INTERVENTIONS:
Drug: GEN1286 — Specified dose on specified days.

SUMMARY:
The purpose of this trial is to evaluate the safety, tolerability, pharmacokinetics (PK), anti-tumor activity and immunogenic potential of GEN1286 in participants with advanced solid tumors.

This trial consists of 2 parts:

* Part A: Dose escalation and dose level expansion
* Part B: Tumor-specific expansion with dose optimization

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must be ≥ 18 years of age at the time of informed consent; have measurable disease according to RECIST 1.1; Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1; adequate organ, bone marrow, liver, coagulation, and renal function; and be willing to provide a pretreatment tumor specimen.
* All participants must have pathologically confirmed diagnosis of advanced solid tumor.
* Participants must have metastatic or unresectable locally advanced, recurrent disease not amenable to further local therapy and must have previously received therapies known to confer clinical benefit (unless ineligible to receive, refused to receive, or therapy is unavailable in the region).

Key Exclusion Criteria:

- Prior treatment with topoisomerase 1-based antibody-drug conjugate (ADC) therapy.

Note: Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2028-05-29 (Estimated); Study Completion 2028-06-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | From first dose until 12 months post last dose of study drug or withdrawal of consent, death, or study closure, whichever occurs first (Up to approximately 3 years 9 months)
Number of Participants With Dose Limiting Toxicities (DLTs) | During first cycle (Cycle length=21 days)
  Toxicities will be graded for severity according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria version 5.0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 3 years 9 months
  ORR is defined as the percentage of participants achieving a partial response (PR) or complete response (CR) as assessed by the investigator based on response evaluation criteria in solid tumors (RECIST) version 1.1.
Disease Control Rate (DCR) | Up to approximately 3 years 9 months
  DCR is defined as the percentage of participants with stable disease (SD) or achieving a PR or CR based on RECIST version 1.1 as assessed by the investigator.
Progression Free Survival (PFS) | Up to approximately 3 years 9 months
  PFS is defined as the time from the start of any treatment to the date of the first documented progression or death due to any cause, whichever occurs first based on RECIST version 1.1 as assessed by the investigator.
Duration of Objective Response (DOR) | Up to approximately 3 years 9 months
  DOR is defined as the time from the first documentation of an objective tumor response (CR or PR) to the first documentation of tumor progression or to death due to any cause, whichever comes first based on RECIST version 1.1 as assessed by the investigator.
Area Under the Plasma or Serum Concentration Time Curve (AUC) of GEN1286 Related Analytes- Antibody-Conjugated Exatecan, Total Antibody (Tab) and u-Exatecan | Predose and postdose at multiple timepoints at end of each cycle, up to approximately 2 years 9 months (Cycle length=21 days)
Maximum Observed Plasma or Serum Concentration (Cmax) of GEN1286 Related Analytes- Antibody-Conjugated Exatecan, Tab and u-Exatecan | Predose and postdose at multiple timepoints at end of each cycle, up to approximately 2 years 9 months (Cycle length=21 days)
Time to Reach Cmax (Tmax) of GEN1286 Related Analytes- Antibody-Conjugated Exatecan, Tab and u-Exatecan | Predose and postdose at multiple timepoints at end of each cycle, up to approximately 2 years 9 months (Cycle length=21 days)
Apparent Terminal Half-life (t1/2) of GEN1286 Related Analytes- Antibody-Conjugated Exatecan, Tab and u-Exatecan | Predose and postdose at multiple timepoints at end of each cycle, up to approximately 2 years 9 months (Cycle length=21 days)
Clearance (CL) of GEN1286 Related Analytes- Antibody-conjugated Exatecan, Tab and u-Exatecan | Predose and postdose at multiple timepoints at end of each cycle, up to approximately 2 years 9 months (Cycle length=21 days)
Volume of Distribution (Vz) of GEN1286 Related Analytes- Antibody-conjugated Exatecan, Tab and u-Exatecan | Predose and postdose at multiple timepoints at end of each cycle, up to approximately 2 years 9 months (Cycle length=21 days)
Trough Concentrations (Ctrough) of GEN1286 Related Analytes- Antibody-conjugated Exatecan, Tab and u-Exatecan | Predose and postdose at multiple timepoints at end of each cycle, up to approximately 2 years 9 months (Cycle length=21 days)
Number of Participants with Antidrug Antibodies (ADA) to GEN1286 | Up to approximately 2 years 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - START San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No